CLINICAL TRIAL: NCT01363648
Title: A Randomized, Double-blind, Placebo-controlled Phase IV Trial for an Evaluation of the Efficacy of Gliatiline® on Post-stroke Patients With Vascular Cognitive Impairment no Dementia
Brief Title: The Efficacy of Gliatiline® on Post-stroke Patients With Vascular Cognitive Impairment no Dementia
Acronym: GLITTER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Joon Bae, Proffessor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLITTER-DW400; MOON KU HAN (Registry Identifier: GLITTER)
Record Dates: First submitted 2011-05-29; First posted 2011-06-01 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Cognitive Impairment; Stroke
Keywords: VCI-HS; stroke; choline alphoscerate
MeSH Terms: conditions — Cognitive Dysfunction; Stroke | interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Choline alfoscerate (Experimental): choline alfoscerate 400mg, 3 times a day, for 12 weeks.
  Interventions: Drug: choline alfoscerate
- placebo (for choline alfoscerate ) (Placebo Comparator): placebo tablet, 3 times a day, for 12 weeks.
  Interventions: Drug: placebo (for choline alphoscerate)

INTERVENTIONS:
Drug: choline alfoscerate — Participants were randomly assigned to twice-daily doses of 400mg choline alphoscerate (alpha-glyceryl phosphoryl choline, Gliatilin®)
  Other Names: Gliatilin®
  Arms: Choline alfoscerate
Drug: placebo (for choline alphoscerate) — Pill manufactured to mimic choline alfoscerate 400mg tablet
  Other Names: placebo
  Arms: placebo (for choline alfoscerate )

SUMMARY:
To date, there are no approved treatments for vascular cognitive impairment (VCI) and the main therapeutic efforts are aimed at controlling vascular risk factors for countering VCI development or progression. Several studies have reported cholinergic deficits in brain and cerebrospinal fluid of patients with VCI. The effect of choline alphoscerate in clinical studies of Alzheimer's disease and VCI improved memory and attention impairments. The purpose of our study is to determine effectiveness of choline alphoscerate vs placebo in improving cognition in post-stroke patients with VCI-non dementia (VCI-ND).

DETAILED DESCRIPTION:
Impaired brain cholinergic neurotransmission has a key role in the deterioration of cognitive functions in Alzheimer's disease and vascular cognitive impairment (VCI). These deficits, although are of different degree than those found in Alzheimer's disease, were suggested to be associated with VCI.To date, there are no approved treatments for vascular dementia(VaD)and the main therapeutic efforts in this field are aimed at controlling vascular risk factors for countering VaD development or progression.

There have also been several trials of cholinesterase inhibitors for treatment of VCI. Available data suggest some evidence of benefit of cholinesterase inhibitors in subcortical vascular dementia and vascular cognitive impairment.

Treated patients had modest benefits in cognition, attention, executive functioning and ability to perform instrumental activities of daily living, but the effect is too limited due to the small numbers of subjects examined and it is complex to establish the clinical relevance of these effects. The majority of clinical studies available on the effect of choline alphoscerate in neurodegenerative and cerebrovascular disorders were reviewed. A comparison of Alzheimer's disease assessment scale-cognitive subscale(ADAS-Cog)analysis with the results obtained on the same item in 4 trials with the cholinesterase inhibitor revealed a more positive trend with the cholinergic precursor choline alphoscerate than with this cholinesterase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients were outpatients (age 25 to 84 years) with vascular cognitive impairment that does not fulfill dementia criteria (vascular cognitive impairment, no dementia(CIND)), had been stroke free for 90 days, together with clinical and radiological evidence of stroke and can perform K-TMT-e A. Cognitive impairment did not meet the Diagnostic and Statistical Manual of Mental Disorders, Revised Third Edition (DSM-III-R) criteria for dementia (ie, they did not have both memory impairment and other cognitive impairment that caused functional deficits).

Exclusion Criteria:

* Exclusion criteria included clinical or radiological evidence of neurodegenerative disorders other than VCI. Patients with major depression or other psychiatric disorders (according to criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) were excluded. Patients who had experienced a myocardial infarction within 3 months of enrollment were excluded (although these patients could be reconsidered for inclusion once 3 months had elapsed), as were those with clinically relevant hepatic, pulmonary, gastrointestinal, or life-threatening disease. Additional reasons for exclusion included pregnancy, a history of alcohol or drug abuse, and contraindications for MRI studies. Medications that affect the cognitive function were not permitted within the last 30 days. Patients were not permitted to receive anticholinergic drugs or cholinergic agents other than gliatilin during the study period.

Ages: 25 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the change of K-TMT-e A of K-VCIHS-NP in the choline alfoscerate vs the placebo groups. | 12 weeks after taking drugs
  Primary analysis compares the change of K-TMT-e A of K-VCIHS-NP from the study entry 12 weeks later in the choline alfoscerate vs the placebo groups.

SECONDARY OUTCOMES:
the change of other determinants of K-VCIHS-NP in the choline alfoscerate vs the placebo groups | 12 weeks after taking drugs
  secondary analysis compares the change of other determinants of K-VCIHS-NP from the study entry 12 weeks later in the choline alfoscerate vs the placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-JOON BAE, Proffessor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang, Seongnam, Gyeoinggido, South Korea

REFERENCES:
- [Background] Parnetti L, Mignini F, Tomassoni D, Traini E, Amenta F. Cholinergic precursors in the treatment of cognitive impairment of vascular origin: ineffective approaches or need for re-evaluation? J Neurol Sci. 2007 Jun 15;257(1-2):264-9. doi: 10.1016/j.jns.2007.01.043. Epub 2007 Feb 28. PMID 17331541